CLINICAL TRIAL: NCT03341754
Title: A Phase 1 Trial With Controlled Human Malaria Infection to Evaluate the Safety, Immunogenicity, and Protective Efficacy of Two-Antigen and Three-Antigen Plasmodium Falciparum DNA Prime-Adenovirus Boost Malaria Vaccine Regimens in Healthy Malaria Naïve Adults
Brief Title: Trial to Evaluate the Safety, Immunogenicity, and Efficacy of Malaria Infection in Malaria Naïve Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: U.S. Army Medical Research and Development Command (U.S. Federal Agency)
Collaborators: University of Oxford (Other); Walter Reed Army Institute of Research (WRAIR) (U.S. Federal Agency); United States Agency for International Development (USAID) (U.S. Federal Agency); Naval Medical Research Center (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: S-14-07; NMRC.2016.0006 (Other: NMRC); NavOx (Other: Sponsor)
Record Dates: First submitted 2017-10-12; First posted 2017-11-14 (Actual); Last update posted 2020-05-06 (Actual); Status verified 2020-05

CONDITIONS: Malaria
Keywords: Malaria Infection
MeSH Terms: conditions — Malaria | interventions — Population Groups

STUDY DESIGN:
Intervention Model Description: The study will include 2 vaccine groups and an infectivity control (IC) group consisting of non-immunized subjects.
Who Masked: Participant
Masking Description: Trial subjects will be blinded from their treatment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Group 1 (D/ChAd63-CA) (Experimental): (2-antigen): 3 doses at 4 week intervals (Week 0, 4, and 8) of DNA prime with D-C + D-A at 2 mg total (1 mg per construct) per dose as two 1 mL IM injections of the blended D-CA, one in each arm, via Biojector 2000 needle-free injection device or an equivalent disposable syringe needle-free injection device. This will be followed after 16 weeks (Week 24) by 1 dose of ChAd63-C + ChAd63-A boost, at a total dose of 1 x 1011 virus particles (vp) (5 x 1010 vp/construct) as a single IM injection of 0.65mL, using a needle and syringe.
  Week 0 = Prime with D-CA Week 4 = Prime with D-CA Week 8 = Prime with D-CA Week 24 = Boost with ChAd63-CA Week 28 = Controlled Human Malaria Infection (CHMI)
  Interventions: Biological: D/ChAd63-CA
- Group 2 (D/ChAd63-CAT) (Experimental): (3-antigen): 3 doses at 4 week intervals (Week 0, 4, and 8) of DNA prime with D-C + D-A + D-T at 3 mg total (1 mg per construct) per dose as two 1 mL intramuscular (IM) injections of the blended D-CAT, one in each arm, via Biojector 2000 needle-free injection device or an equivalent disposable syringe needle-free injection device. This will be followed after 16 weeks (Week 24) by 1 dose of ChAd63-C + ChAd63-A + ChAd63-T boost, at a total dose of 1.5 x 1011 vp (5 x 1010 vp/construct) as a single IM injection of 1.0mL, using a needle and syringe.
  Week 0 = Prime with D-CAT Week 4 = Prime with D-CAT Week 8 = Prime with D-CAT Week 24 = Boost with ChAd63-CAT Week 28 = Controlled Human Malaria Infection (CHMI)
  Interventions: Biological: D/ChAd63-CAT
- Infectivity Control (IC) (Active Comparator): Subjects will be exposed to the bites of 5 Anopheles stephensi mosquitoes carrying infectious Pf sporozoites within a controlled clinical environment.
  Week 28 = Controlled Human Malaria Infection (CHMI)
  Interventions: Other: Infectivity Control (IC) Group

INTERVENTIONS:
Biological: D/ChAd63-CA — Priming Component (DNA) = NMRC-M3V-D-PfCA (D-CA) Vaccine Boosting Component = ChAd63-PfCA
  Arms: Group 1 (D/ChAd63-CA)
Biological: D/ChAd63-CAT — Priming Component (DNA) = NMRC-M3V-D-PfCAT (D-CAT) Boosting Component = ChAd63-PfCAT
  Arms: Group 2 (D/ChAd63-CAT)
Other: Infectivity Control (IC) Group — Subjects will be exposed to bites of 5 Anopheles stephensi mosquitoes carrying infectious Pf sporozoites within a controlled clinical environment.
  Other Names: Controlled Human Malaria Infection (CHMI)
  Arms: Infectivity Control (IC)

SUMMARY:
This is a study designed to assess the safety, tolerability, immunogenicity, and protective efficacy of 2 heterologous prime-boost vaccine regimens in healthy, malaria naïve adults. The study will include 2 vaccine groups and an infectivity control (IC) group consisting of non-immunized subjects. Subjects to be immunized will be randomly assigned to one of two vaccine groups.

DETAILED DESCRIPTION:
This is a study designed to assess the safety, tolerability, immunogenicity, and protective efficacy of 2 heterologous prime-boost vaccine regimens in healthy, malaria naïve adults. The study will include 2 vaccine groups and an infectivity control (IC) group consisting of non-immunized subjects. Subjects to be immunized will be randomly assigned to one of two vaccine groups. Approximately 4 weeks after administration of the boosting immunization the vaccinated groups and the IC group will participate in CHMI wherein subjects will be exposed to the bites of 5 Anopheles stephensi mosquitoes carrying infectious Pf sporozoites within a controlled clinical environment. Protection will be determined by the examination of thick blood smears through 28 days post-CHMI and by retrospective PCR analysis for the presence of blood stage parasites. All groups will be enrolled and evaluated in one cohort. Due to a limit in the number of subjects who can undergo malaria challenge at the facility in one day, CHMI will be conducted over two days.

Group 1 (2-antigen): 3 doses at 4 week intervals (Week 0, 4, and 8) of DNA prime with D-C + D-A at 2 mg total (1 mg per construct) per dose as two 1 mL IM injections of the blended D-CA, one in each arm, via Biojector 2000 needle-free injection device or an equivalent disposable syringe needle-free injection device. This will be followed after 16 weeks (Week 24) by 1 dose of ChAd63-C + ChAd63-A boost, at a total dose of 1 x 1011 virus particles (vp) (5 x 1010 vp/construct) as a single IM injection of 0.65mL, using a needle and syringe.

Group 2 (3-antigen): 3 doses at 4 week intervals (Week 0, 4, and 8) of DNA prime with D-C + D-A + D-T at 3 mg total (1 mg per construct) per dose as two 1 mL intramuscular (IM) injections of the blended D-CAT, one in each arm, via Biojector 2000 needle-free injection device or an equivalent disposable syringe needle-freeinjection device. This will be followed after 16 weeks (Week 24) by 1 dose of ChAd63-C + ChAd63-A + ChAd63-T boost, at a total dose of 1.5 x 1011 vp (5 x 1010 vp/construct) as a single IM injection of 1.0mL, using a needle and syringe.

ELIGIBILITY:
Inclusion Criteria:

* Adults (male or non-lactating, non-pregnant female) between 18 to 50 years of age at the time of enrollment
* Available and willing to participate for duration of study
* Able and willing to provide a written informed consent
* Able to complete an Assessment of Understanding (Appendix C) with a score of at least 80% correct
* In good general health with no clinically significant health problems as established by medical history, physical examination, and laboratory screening
* Men and women of childbearing potential must agree to consistently use effective means of birth control throughout the duration of the study
* Sexually active females, unless surgically sterile or at least 1 year postmenopausal, must use an effective method of avoiding pregnancy (including oral or implanted contraceptives, intrauterine device, female condom, diaphragm with spermicide, cervical cap, abstinence, use of a condom by the sexual partner or sterile sexual partner) from 14 days prior to the first immunization and must agree to continue using such precautions during the study and for 6 months after the last study visit (which occurs at 90 days after CHMI).
* If female subjects are unable to bear children due to menopause or have had a procedure performed (tubal ligation or hysterectomy), a medical note from a physician is required.
* If post-menopausal, subjects must have experienced at least 1 year of amenorrhea and provide a medical note from her physician documenting this medical history.
* Sexually active men must agree to use effective means of birth control such as barrier methods (use of a condom) from the day of the first immunization and for the duration of the study (through 3 months after CHMI). Vasectomy is considered an adequate means of birth control. Men who underwent sterilization or vasectomy must provide a medical note from his physician documenting such procedure.
* Agree not to travel to a malaria endemic area during the course of the study
* Agree to refrain from blood donation during the study and for 3 years following CHMI
* Must be willing to take anti-malarial treatment after CHMI, if indicated.
* Must agree to stay in a pre-determined hotel near the NMRC CTC during the designated post-CHMI followup period from approximately 7 days after malaria challenge until antimalarial treatment is completed, if indicated

Exclusion Criteria:

* Weight < 110 pounds
* Body mass index (BMI) > 35 kg/m2
* Pregnant (positive urine pregnancy test) or nursing at screening or plans to become pregnant or nurse at any period from the time of enrollment through 6 months after the last study visit (which will occur at 90 days after CHMI).
* Receipt of any investigational malaria vaccine
* Any history of malaria infection
* Travel to a malaria endemic region within 6 months of enrollment or during the study (from enrollment through 3 months after CHMI)
* History of long-term residence (>5 years) in an area known to have significant transmission of P falciparum (http://www.cdc.gov/malaria/map/)
* History of clinically significant contact dermatitis or sensitivity to products that contain Kathon, such as shampoos, conditioners, soaps, detergents, moisturizers, lotions, baby wipes, or cosmetics
* Positive CSP and AMA1 ELISpot assay at screening
* Positive CSP and AMA1 ELISA assay at screening
* Seropositive for the human immunodeficiency virus (HIV), hepatitis C virus (HCV), and/ or hepatitis B surface antigen (HBsAg)
* Positive sickle cell screening test, including evidence of sickle cell trait or sickle cell anemia (due to its effect on subject's susceptibility to malaria)
* History of thalassemia or thalassemia trait (due to its effect on subject's susceptibility to malaria)
* Participation in any clinical study involving another investigational vaccine, drug, or other products within 60 days prior to the first immunization or plan to participate in such a clinical study during or within 1 month following the active study phase of the study (from the day of the first immunization through 3 months after CHMI)
* Allergy to any component of the vaccine formulation or serious adverse reaction to other vaccines (such as hives, anaphylaxis, respiratory difficulty, angioedema, or abdominal pain)
* History of a severe and/or anaphylactic response to mosquito-bites
* Known allergy to chloroquine phosphate, atovaquone/proguanil, or artemether/lumefantrine, which will be used to treat subjects who may develop malaria after Plasmodium falciparum challenge
* History of psoriasis (given its interaction with chloroquine)
* History of porphyria
* History of hemolytic anemia
* Use or planned use of any drugs with significant anti-malarial activity, such as doxycycline, clindamycin, azithromycin, or trimethoprim/sulfamethoxazole among others that would coincide with periods of CHMI or post-CHMI followup
* Has evidence of increased cardiovascular disease risk (> 5%-10%, 5-year risk)
* As determined by the method of Gaziano et al (2008, Appendix D)
* Risk factors include sex, age (years), smoking status, body mass index (BMI, kg/m2), presence or absence of diabetes mellitus, and blood pressure.
* An abnormal EKG, defined as one showing Q waves and/or significant ST-T wave changes, left ventricular hypertrophy, any non-sinus rhythm (excluding isolated premature atrial contraction), right or left bundle branch block, or advanced (secondary or tertiary) A-V heart block
* Current or chronic use of systemic immunosuppressant pharmacotherapy or immunomodulators; however, subjects may be allowed to use inhaled steroids or topical steroids.
* History of splenectomy (given its effects on immunity to malaria)
* Receipt of immunoglobulins and/or any blood products within 90 days of scheduled immunization
* History of neurologic disorder (including seizures or migraine headache)
* History of cancer (except for basal cell carcinoma of the skin)
* Current significant medical condition (cardiovascular, pulmonary, hepatic, renal, or hematological) or evidence of any other serious underlying medical condition identified by medical history, physical examination, or laboratory screening tests
* History of any other illness or condition which, in the investigator's judgment, may substantially increase the risk associated with the subject's participation in the protocol or compromise the scientific objectives. This may include psychiatric disorders (such as personality disorders, anxiety disorders, major depressive disorder or schizophrenia) or behavioral tendencies (including active alcohol or drug abuse) discovered during the screening process that in the opinion of the investigator would make compliance with the protocol difficult
* Plan for surgery during the study (from enrollment until 3 months post-CHMI) with the exception of minor cutaneous procedures
* Females who are pregnant or nursing, or plan to become pregnant or nurse during the study period (from enrollment through 3 months post CHMI) or within 6 months after the last study visit
* Any other significant finding that in the opinion of the investigator would increase the risk of having an adverse outcome from participating in this study or compromise the scientific objectives

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 52 (Actual)
Dates: Start 2018-09-15 (Actual); Primary Completion 2019-10-28 (Actual); Study Completion 2020-03-23 (Actual)

PRIMARY OUTCOMES:
Occurrence of Serious Adverse Events | Through day 7 after each immunization
  Occurrence of Serious Adverse Events following immunization through day 7 after each immunization
Occurrence of Abnormal Physical Symptoms (Clinical Abnormalities) | Through day 28 after each immunization
  Occurrence of Abnormal Physical Findings following immunization through day 28 after each immunization.
  Grading Scale:
  Grade 1= No interference with activity; Grade 2= Some interference with activity; Grade 3=Prevents daily activity; Grade 4= ER visit or hospitalization
Occurrence of Abnormal Laboratory Values | Through day 28 after each immunization
  Occurrence of Abnormal Laboratory Values following immunization through day 28 after each immunization
Occurrence of Any Serious Adverse Events Throughout the Study Period | Enrollment through 3 months after CHMI
  Occurrence of Any Serious Adverse Events Throughout the Study Period, from enrollment through 3 months after CHMI

SECONDARY OUTCOMES:
Vaccine Efficacy Determined by Time to Development of Parasitemia | after CHMI: Days 7 - 28
  Vaccine Efficacy Determined by Time to Development of Parasitemia as measured by microscopic examination of thick smears and by Polymerase Chain Reaction (PCR) after CHMI and PCR analysis conducted retrospectively
Measurement of Antibody Titers Against Sporozoite and Erythrocyte Stage Parasites | Days 231 and 286
  Measurement of antibody titers against sporozoite and erythrocyte stage parasites by immunofluorescence assay (IFA) using sera/plasma
Measure of correlation between pre-immunization HuAd5 neutralizing antibody titers and the protective efficacy against CHMI and humoral and cellular immune responses of the 2 prime-boost regimens | HuAd5: Days -14 to -1; Cellular Immunity: Days -14 to -1, 84, 168 and 195; Humoral Immunity: Days -14 to -1, 14, 28, 42, 56, 70, 84, 168, 195
  Assess the association between the subjects' pre-immunization neutralizing antibody titers to HuAd5 and the protective efficacy and humoral and cellular immunogenicity, of these prime-boost regimens to CSP, AMA1 and TRAP as measured by ELISA and FluoroSpot assays
Comparison of Immunogenicity of the 2 Vaccine Regimens | Days 1 - 286
  Comparison of immunogenicity,of the 2 heterologous prime-boost vaccine regimens (D/ChAd63-CA vs. D/ChAd63-CAT

CONTACTS AND LOCATIONS:
Overall Officials: Nimfa Teneza-Mora, MD, Principal Investigator — United States Military Malaria Vaccine Program, NMRC
Locations (2):
- United States (2):
  - NMRC Clinical Trials Center, Bethesda, Maryland
  - WRAIR, Silver Spring, Maryland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Beadle C, Hoffman SL. History of malaria in the United States Naval Forces at war: World War I through the Vietnam conflict. Clin Infect Dis. 1993 Feb;16(2):320-9. doi: 10.1093/clind/16.2.320. PMID 8443317
- [Background] Breman JG, Alilio MS, Mills A. Conquering the intolerable burden of malaria: what's new, what's needed: a summary. Am J Trop Med Hyg. 2004 Aug;71(2 Suppl):1-15. PMID 15331814
- [Background] Buchbinder SP, Mehrotra DV, Duerr A, Fitzgerald DW, Mogg R, Li D, Gilbert PB, Lama JR, Marmor M, Del Rio C, McElrath MJ, Casimiro DR, Gottesdiener KM, Chodakewitz JA, Corey L, Robertson MN; Step Study Protocol Team. Efficacy assessment of a cell-mediated immunity HIV-1 vaccine (the Step Study): a double-blind, randomised, placebo-controlled, test-of-concept trial. Lancet. 2008 Nov 29;372(9653):1881-1893. doi: 10.1016/S0140-6736(08)61591-3. Epub 2008 Nov 13. PMID 19012954
- [Background] Epstein JE, Rao S, Williams F, Freilich D, Luke T, Sedegah M, de la Vega P, Sacci J, Richie TL, Hoffman SL. Safety and clinical outcome of experimental challenge of human volunteers with Plasmodium falciparum-infected mosquitoes: an update. J Infect Dis. 2007 Jul 1;196(1):145-54. doi: 10.1086/518510. Epub 2007 May 29. PMID 17538895
- [Background] Ogwang C, Afolabi M, Kimani D, Jagne YJ, Sheehy SH, Bliss CM, Duncan CJ, Collins KA, Garcia Knight MA, Kimani E, Anagnostou NA, Berrie E, Moyle S, Gilbert SC, Spencer AJ, Soipei P, Mueller J, Okebe J, Colloca S, Cortese R, Viebig NK, Roberts R, Gantlett K, Lawrie AM, Nicosia A, Imoukhuede EB, Bejon P, Urban BC, Flanagan KL, Ewer KJ, Chilengi R, Hill AV, Bojang K. Safety and immunogenicity of heterologous prime-boost immunisation with Plasmodium falciparum malaria candidate vaccines, ChAd63 ME-TRAP and MVA ME-TRAP, in healthy Gambian and Kenyan adults. PLoS One. 2013;8(3):e57726. doi: 10.1371/journal.pone.0057726. Epub 2013 Mar 19. PMID 23526949
- [Background] Roestenberg M, O'Hara GA, Duncan CJ, Epstein JE, Edwards NJ, Scholzen A, van der Ven AJ, Hermsen CC, Hill AV, Sauerwein RW. Comparison of clinical and parasitological data from controlled human malaria infection trials. PLoS One. 2012;7(6):e38434. doi: 10.1371/journal.pone.0038434. Epub 2012 Jun 11. PMID 22701640
- [Background] Verhage DF, Telgt DS, Bousema JT, Hermsen CC, van Gemert GJ, van der Meer JW, Sauerwein RW. Clinical outcome of experimental human malaria induced by Plasmodium falciparum-infected mosquitoes. Neth J Med. 2005 Feb;63(2):52-8. PMID 15768480